CLINICAL TRIAL: NCT00404924
Title: A Phase III Study to Assess the Efficacy of ZD6474 (ZACTIMA™) Plus Best Supportive Care Versus Best Supportive Care in Patients With Locally Advanced or Metastatic (Stage IIIB-IV) Non-Small Cell Lung Cancer After Therapy With an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR TKI)
Brief Title: ZD6474 (ZACTIMA™) Phase III Study in EGFR Failures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00044; EUDRACT Number 2006-002384-12
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non-Small-Cell Lung Carcinoma; Adenocarcinoma; Squamous Cell Carcinoma; Large Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Squamous Cell; Carcinoma, Large Cell | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator): Best Supportive Care
  Interventions: Other: Best Supportive Care
- 2 (Experimental): Vandetanib + Best Supportive Care
  Interventions: Drug: ZD6474 (vandetanib); Other: Best Supportive Care

INTERVENTIONS:
Drug: ZD6474 (vandetanib) — once daily oral tablet
  Other Names: ZACTIMA™
  Arms: 2
Other: Best Supportive Care — standard of care

SUMMARY:
This study is being carried out to assess if adding ZD6474 to best supportive care (BSC) is more effective than best supportive care alone, for the treatment of patients with non-small cell lung cancer, whose disease has recurred after previous chemotherapy and an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR TKI). ZD6474 is a new anti-cancer drug in development that works in a different way to standard chemotherapy drugs. It targets the growth of new blood vessels to a tumour and thereby might slow the rate at which the tumour may grow. Early studies indicate that ZD6474 has a positive effect on the time that a tumour may take to progress to a further stage. Approximately 930 patients will take part in this study. It will be conducted in hospitals and clinics in North and South America, Europe and Asia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Non-small cell lung cancer for which the standard cancer treatments of surgery, chemotherapy, radiation or other anticancer drugs are no longer appropriate treatments for you.

Exclusion Criteria:

* Patients who have had standard cancer treatments of surgery, chemotherapy or other systemic anti-cancer therapy within 4 weeks before start of study therapy.
* Three or more prior chemotherapy regimens.
* Significant cardiovascular events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140 (Actual)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (102):
- United States (2):
  - Research Site, Tucson, Arizona
  - Research Site, Germantown, Tennessee
- Argentina (6):
  - Research Site, Bahía Blanca
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Australia (5):
  - Research Site, Fitzroy
  - Research Site, Perth
  - Research Site, St Leonards
  - Research Site, Tugan
  - Research Site, Woodville South
- Austria (3):
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (7):
  - Research Site, Antwerp
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (8):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Xi'an
- France (7):
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Pierre-Bénite
  - Research Site, Toulon Armees
- Germany (12):
  - Research Site, Bad Berka
  - Research Site, Donaustauf
  - Research Site, Frankfurt
  - Research Site, Gauting
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Karlsruhe
  - Research Site, Leipzig
  - Research Site, Löwenstein
  - Research Site, Mannheim
  - Research Site, München
- Research Site, Hong Kong, Hong Kong
- Israel (4):
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Tel Litwinsky
  - Research Site, Ẕerifin
- Italy (12):
  - Research Site, Ancona
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, S.Andrea Delle Fratte
  - Research Site, Sondalo
  - Research Site, Udine
- Mexico (2):
  - Research Site, México
  - Research Site, Zapopan
- Research Site, Saint Maartenskliniek, Netherlands
- Research Site, Lima, Peru
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Manila
  - Research Site, Quezon City
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Seongnam
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (4):
  - Research Site, Baracaldo(Vizcaya)
  - Research Site, Barcelona
  - Research Site, Santander
  - Research Site, Valencia
- Taiwan (7):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Kaohsiung Hsien
  - Research Site, Liou Ying Township
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, Chelmsford
  - Research Site, Dundee
  - Research Site, Maidstone
  - Research Site, Manchester

REFERENCES:
- [Derived] Platt A, Morten J, Ji Q, Elvin P, Womack C, Su X, Donald E, Gray N, Read J, Bigley G, Blockley L, Cresswell C, Dale A, Davies A, Zhang T, Fan S, Fu H, Gladwin A, Harrod G, Stevens J, Williams V, Ye Q, Zheng L, de Boer R, Herbst RS, Lee JS, Vasselli J. A retrospective analysis of RET translocation, gene copy number gain and expression in NSCLC patients treated with vandetanib in four randomized Phase III studies. BMC Cancer. 2015 Mar 23;15:171. doi: 10.1186/s12885-015-1146-8. PMID 25881079
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=342&filename=CSR-D4200C00044.pdf
- See also: CSR-D4200C00044.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=342&filename=CSR-D4200C00044.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 08 November 2006, last patient enrolled 09 October 2008, cut off date 19 October 2009. 1168 patients were enrolled in the study.
Groups:
- Vandetanib 300 mg: vandetanib (300 mg daily) plus best supportive care
- Placebo: Placebo plus best supportive care
Period: Overall Study
Arm/Group | Vandetanib 300 mg | Placebo
Started | 617 (randomised patients) | 307 (randomised patients)
Completed | 14 (ongoing study treatment at data cut-off) | 1 (ongoing study treatment at data cut-off)
Not Completed | 603 | 306
Not completed — Adverse Event | 75 | 16
Not completed — Condition under investigation worsened | 475 | 264
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 26 | 13
Not completed — Other | 25 | 11
Not completed — Randomised but not received treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib 300 mg | Placebo | Total
Number analyzed (Participants) | 617 | 307 | 924
Age, Continuous [Mean (Full Range); unit: years] | 59.8 [20 to 85] | 60.6 [21 to 84] | 60 [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329 | 160 | 489
  Male | 288 | 147 | 435

OUTCOME MEASURES:

1. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median time (in months) from randomisation until objective disease progression (determined by RECIST assessments) or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable RECIST assessment
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomisation until objective disease progression
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 617 | 307
month | 1.9 [1.84 to 2.23] | 1.8 [1.74 to 1.84]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the number of patients that are responders ie those patients with a confirmed best objective response of complete response (CR) or partial response (PR) as defined by RECIST criteria.
  The categories for best objective response are CR, PR, stable disease (SD)>= 8 weeks, progressive disease (PD) or NE.
Time Frame: Each patient was assessed for objective response from the sequence of RECIST scan data up to data cut off. RECIST tumour assessments carried out every 8 weeks from randomisation until objective disease progression.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 617 | 307
Participants | 16 | 2

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is defined as the number of patients who achieved disease control at 8 weeks following randomisation. Disease control at 8 weeks is defined as a best objective response of complete response (CR), partial response (PR) or stable disease (SD) >= 8 weeks
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomisation until objective disease progression
Measure: Number; unit: Participants
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 617 | 307
Participants | 189 | 48

4. Secondary Outcome: Duration of Response (DoR)
Description: Response is defined as a confirmed best objective response of CR or PR. Duration of response is defined as time from the date of first documented response until date of documented progression or death in the absence of disease progression (provided death is within 3 months of last RECIST assessment)
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomisation until objective disease progression
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 16 | 2
Weeks | 23.9 [16.57 to 27.00] | 24.3 [16.00 to 32.57]

5. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from date of randomization until death. Any blinded/unknown patient which have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive (ie, their status must be known at the censored date and should not be lost to follow up or unknown).
Time Frame: Time to death in months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 617 | 307
Months | 8.5 [7.81 to 9.76] | 7.8 [6.08 to 9.17]

6. Secondary Outcome: Time to Deterioration of Disease-related Symptoms (TDS) by Questionnaire - the Lung Cancer Subscale (LCS) a Selection of the FACT-L Focusing on Symptoms of Lung Cancer Plus Pain and Fatigue (LCS-PF)
Description: Time to deterioration in symptoms is defined as the interval from the date of randomization to the first assessment of 'worsened' with no visit assessment of 'improved' within the next 28 days. Where assessment is by a selection of questions from the Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) questionnaire.
Time Frame: Disease-related symptom assessments are to be administered at screening (within 7 days before the first dose of study medication) and every 4 weeks thereafter, at discontinuation of study treatment and at the 30-day follow-up visit
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Vandetanib 300 mg | Placebo
Number analyzed (Participants) | 617 | 307
weeks | 6.1 [5.14 to 8.14] | 7.1 [5.86 to 8.43]

ADVERSE EVENTS:
Description: The Safety Analysis Set included 922 patients (619 vandetanib & 303 placebo), which represents more than 99% of all randomized pts. 2 (1 in each arm) were excluded from the SAS as they were not dosed. Additionally 3 pts randomized to receive placebo received at least one dose of vandetanib, these 3 pts are included in the vandetanib arm in the SAS
Groups:
- Vandetanib: Vandetanib 300 mg
- Placebo: Placebo
Arm/Group | Vandetanib | Placebo
Serious Adverse Events (participants affected / at risk) | 160/619 | 63/303
Other Adverse Events (participants affected / at risk) | 557/619 | 234/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=619) | Placebo (N=303)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Cardiac Failure (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Valve Disease (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0
Visual Acuity Reduced (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 2 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Neutropenic Colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 5 | 1
Death (General disorders) | 3 | 0
Fatigue (General disorders) | 3 | 1
Pyrexia (General disorders) | 3 | 3
Chest Pain (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 1
Cytolytic Hepatitis (Hepatobiliary disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 2 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 21 | 6
Sepsis (Infections and infestations) | 3 | 1
Lung Infection (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Catheter Site Infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridial Infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Injection Site Abscess (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram T Wave Inversion (Injury, poisoning and procedural complications) | 1 | 0
Lipase Increased (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 5 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 3
Cerebral Ischaemia (Nervous system disorders) | 3 | 0
Cerebrovascular Accident (Nervous system disorders) | 3 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Partial Seizures (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 2
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 3 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 0
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Jugular Vein Thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0
Visceral Arterial Ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=619) | Placebo (N=303)
Anaemia (Blood and lymphatic system disorders) | 19 | 19
Diarrhoea (Gastrointestinal disorders) | 284 | 34
Nausea (Gastrointestinal disorders) | 138 | 51
Constipation (Gastrointestinal disorders) | 88 | 63
Vomiting (Gastrointestinal disorders) | 82 | 36
Stomatitis (Gastrointestinal disorders) | 34 | 13
Abdominal Pain (Gastrointestinal disorders) | 26 | 19
Fatigue (General disorders) | 109 | 50
Asthenia (General disorders) | 62 | 30
Pyrexia (General disorders) | 44 | 29
Oedema Peripheral (General disorders) | 33 | 29
Weight Decreased (General disorders) | 47 | 18
Electrocardiogram Qt Prolonged (General disorders) | 37 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 143 | 63
Back Pain (Musculoskeletal and connective tissue disorders) | 54 | 19
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 22 | 20
Dizziness (Nervous system disorders) | 68 | 27
Headache (Nervous system disorders) | 61 | 24
Insomnia (Psychiatric disorders) | 63 | 24
Proteinuria (Renal and urinary disorders) | 56 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 108 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 98 | 52
Rash (Skin and subcutaneous tissue disorders) | 258 | 33
Pruritus (Skin and subcutaneous tissue disorders) | 70 | 16
Dry Skin (Skin and subcutaneous tissue disorders) | 49 | 8
Hypertension (Vascular disorders) | 160 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.